CLINICAL TRIAL: NCT05165927
Title: Comparison of Methods in Post Operative Hip Arthroscopy Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-4753
Record Dates: First submitted 2021-12-03; First posted 2021-12-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hip Injuries
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: ACT's that collect data during visits will be blinded to what group the subject is in to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BFR Group (Experimental): BFR cuffs will be used for specific exercises and added to the current SOC for post hip scope PT.
  Interventions: Device: BFR
- SOC Group (No Intervention): Current SOC for post hip scope PT will be assigned.

INTERVENTIONS:
Device: BFR — BFR cuffs will be used at home during specified exercises in addition to SOC for post hip scope PT.
  Arms: BFR Group

SUMMARY:
The investigators plan to investigate the efficacy of blood flow restriction (BFR) therapy in post operative rehabilitation following hip arthroscopy. BFR has shown to be great at helping the recovery process. SAGA is a well-known smart training technology company, and the investigators aim to partner with SAGA to use the BFR cuffs as the intervention method. The BFR cuff will be added to the current SOC for hip scope PT for the intervention group.

DETAILED DESCRIPTION:
Study Design and Research Methods i. Timeline: Treatment Protocol duration 12 weeks per participant beginning post operative day 1 following hip arthroscopy. PRO's will be collected out to 2 years post-surgery and standard rehabilitation will follow the 12-week intervention period for both the control and experimental group. Study will be a 2-year timeline in total.

ii. Procedures: Patients will be randomized to control group, who will undergo Steadman Hawkins Clinic Denver's standard hip arthroscopy rehab protocol (see appendix) or to the intervention group, who will undergo standard rehab protocol with addition of BFR. Subjects will be randomized 1:1 for intervention vs. control and controlled for gender assigned at birth.

iii. Frequency of BFR Training: 6 days per week phase 1, 3 days per week phases 2 and 3 iv. Frequency of clinic visits PT: 1 day per week v. Intervention Group: The following exercises outlined are the specific exercises that will be performed in addition to SOC. Only these exercises will involve the use of the BFR cuff.

1. Phase 1 (post operative weeks 1-3)

   1. Dosage: 80% limb occlusion pressure (LOP). 30x15x15x15 repetitions with 30 sec rests between sets. At least 1 min rest between exercises with occlusion OFF.
   2. Frequency: All 3 exercises performed at least 6 days per week. The first of these sessions will be performed in clinic supervised by PT to assess LOP and form prior to performance at home
   3. Exercises:

   i. Week 1: quadriceps set, gluteal set, hamstring set ii. Week 2: short arc quad, hook lying adduction/internal rotation isometric, hook lying abduction/external rotation isometric iii. Week 3: long arc quad, bridge, standing hamstring curl
2. Phase 2 (weeks 4-6)

   1. Dosage: 80% LOP. 30x15x15x15 repetitions with 30 sec rests between sets. At least 1 min rest between exercises with occlusion OFF
   2. Frequency: All 3 resistive exercises performed at least 3 days per week. The first of these sessions will be performed in clinic supervised by PT to assess LOP and form prior to performance at home
   3. Exercises:

   i. Week 4: mini squat, prone hip extension over plinth, quadruped rock ii. Week 5: mid-range squat, modified single leg bridge foot on ball, heel slide strap assist iii. Week 6: step up, standing hip abduction, single leg bridge
3. Phase 3 (weeks 6-12)

   a. Dosage: 80% LOP at 20-30% 1 RM.1 RM re-evaluated every 2 weeks to adjust resistance prescription. 30x15x15x15 repetitions with 30 sec rests between sets. At least 1 min rest between exercises with occlusion OFF b. Frequency: All 3 resistive exercises performed at least 3 days per week. The first of these sessions will be performed in clinic supervised by PT to assess LOP and form prior to performance at home c. Exercises: i. Weeks 6-12: Single leg squat to 45 deg knee flexion (holding weight as tolerated), single leg Romanian dead lift (holding weight a weight as tolerated), Bulgarian split squat (holding a weight as tolerated)
4. Phase 4 (12+ weeks) a. BFR intervention will be discontinued at 12 weeks and participants will progress per standard protocol for the remainder of their rehabilitation course vi. Control Group

1. Control group will follow the standard of care outlined in Appendix A. vii. Criteria for progression within the BFR specific exercise protocol

1. Regardless of functional performance, patients will not be allowed to progress ahead of the time-based exercise prescription in the BFR protocol. However, if the treating therapist determines that the current week's exercise prescription is too difficult for the patient, subject may return to the prior week's exercise set until able to advance.

ELIGIBILITY:
Inclusion Criteria:

* patients with labral tears, femoroacetabular impingement syndrome, loose bodies, ligamentum teres tears, and related intra-articular pathology to be treated with hip arthroscopy. Patients must also have access to a smartphone device in order to utilize the SAGA BFR application for use. The application is free to use.

Exclusion Criteria:

* bilateral hip surgeries to be performed within 12 weeks of each other, concomitant Peri-acetabular osteotomy, soft tissue repairs (hamstring, glute repairs), clinically diagnosed hip dysplasia, and the following BFR contraindications:

  * Deep Vein Thrombosis (DVT)
  * Pulmonary Embolism
  * Hemorrhagic/Thrombolytic Stroke
  * Clotting Disorders
  * Hemophilia or taking blood thinners
  * Pregnant or up to 6 months post-partum
  * Untreated Hypertension
  * Untreated Hypotension
  * Rhabdomyolysis or recent traumatic injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip extensor strength | 2 Years
  1. Strength of hip extensors via handheld dynamometry (HHD) and reported as a measure of limb symmetry index (LSI) comparing operative limb to non-operative limb. By 3 months post operatively, patients should be approaching 70% LSI in order to safely initiate impact activities such as jogging. Prior to discharge from therapy, patients should achieve at least 90% LSI per standard protocol.

SECONDARY OUTCOMES:
additional hip musculature strength | 2 Years
  1. Strength of hip flexors, abductors and adductors via handheld dynamometry (HHD) and reported as a measure of limb symmetry index (LSI) comparing operative limb to non-operative limb. By 3 months post operatively, patients should be approaching 70% LSI in order to safely initiate impact activities such as jogging. Prior to discharge from therapy, patients should achieve at least 90% LSI per standard protocol.
single leg squat test | 2 Years
  2. Performance on a Repeated Single Leg Squat test to 45 deg knee flexion over the course of 90 seconds reported as a measure of LSI. Prior to initiation of impact activities such as jogging (usually around 3 months), patient should be approaching 70% LSI per standard protocol and 90% by time of discharge.
i-HOT | 2 Years
  Range 0 (poor health) - 100 (good health); MCD = Δ13
LEFS | 2 Years
  Range 0 (extreme difficulty) - 100 (extreme difficulty); MDIC = Δ 123
PROMIS pain | 2 Years
  PROMIS Pain: Range 0 (low pain) - 100 (high pain); MDC = Δ 85.
Brief Resiliency Score | 2 Years
  Range 1 (low resilience) - 5 (high resilience)
PROMIS physical function | 2 Years
  PROMIS Physical Function: Range 0 (low function) - 100 (high function); MDC = Δ 85
range of motion (ROM) | 2 Years
  MDC = Δ low (1-2.99) to normal (3-4.3) to high (4.31-5)
Tegner Activity Scale | 2 Years
  Range 0 (disability because of knee problems) - 10 (national or international level soccer)

CONTACTS AND LOCATIONS:
Overall Officials: James Genuario, MD, Principal Investigator — University of Colorado SOM
Locations (1):
- UCHealth Steadman Hawkins Clinic Denver, Englewood, Colorado, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT05165927/ICF_001.pdf